CLINICAL TRIAL: NCT01583634
Title: Accuracy of Oximeters With Hypoxia and Methemoglobin or Carboxyhemoglobin
Status: Completed | Type: Observational
Sponsor: Mespere Lifesciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MLS STP-9100001
Record Dates: First submitted 2012-04-12; First posted 2012-04-24 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: 9 subjects (male and female)
  Interventions: Device: Mespere Oximeter; Device: Radiometer OSM-3 Co-Oximeter

INTERVENTIONS:
Device: Mespere Oximeter — Mespere oximeter provides non-invasive venous blood oxygen saturation.
Device: Radiometer OSM-3 Co-Oximeter — OSM-3, a Radiometer manufactured hemoximeter, is intended for the photometric determination of hemoglobin.

SUMMARY:
Accuracy of the oximeter.

DETAILED DESCRIPTION:
The conventional pulse oximeter has been a standard in clinical care for non-invasive hemodynamic monitoring, which only measures the arterial blood oxygenation. There are many clinical situations where tissue hypoxia may exist despite normal values obtained by conventional pulse oximeter. This can be cause by inadequate monitoring of oxygen demand (i.e. venous oxygen saturation) of the tissues.

The existing method for venous blood oxygenation monitored is either through an invasive fiber optic catheter, or intermittently by blood sampling and CO-oximetry. However, catheterization can be costly and can include inherent risks. Therefore, due to the inherent risks of catheterization, venous oximetry is limited only to those critically ill patients. The clinical application of venous oximetry is numerous, including severe sepsis and septic shock, severe trauma and hemorrhagic shock, and heart failure and cardiac arrest.

More complete information on patient hemodynamics can be provided by non-invasively monitoring of venous blood oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 21 and 49 years of either gender

Exclusion Criteria:

* smokers
* pregnancy
* any chronic medical condition including heart disease, hypertension, pulmonary disease, liver or kidney disease
* obesity
* evidence of abnormal neck vein anatomy

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers between the ages of 21 and 49 years of either gender, and a range of skin tones
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Venous Oxygen Saturation Accuracy Verification against Co-Oximeter | approximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Induced Hypoxia Lab, San Francisco, California, United States